CLINICAL TRIAL: NCT03459794
Title: The Effects of Ivermectin on Human Innate Immunity Against Filarial Parasites
Brief Title: Ivermectin and Human Immunity
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Georgia (Other)
Responsible Party: Principal Investigator, Adrian Wolstenholme, Professor, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: STUDY00005069
Record Dates: First submitted 2018-02-22; First posted 2018-03-09 (Actual); Results first posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-04

CONDITIONS: Ivermectin
MeSH Terms: interventions — Ivermectin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ivermectin (Active Comparator): Ivermectin will be administered once at 150mcg/kg, orally.
  Interventions: Drug: Ivermectin
- Control (Placebo Comparator): An oral placebo will be administered once
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ivermectin — 150 mcg/kg ivermectin, by mouth.
  Arms: Ivermectin
Other: Placebo — An oral placebo will be administered, once
  Arms: Control

SUMMARY:
We hypothesize that ivermectin, a drug used to treat parasitic worm infections, interacts with the human innate immune system and that this contributes to its anti-parasitic effects. Participants will donate blood before and after being administered the normal human dose of the drug. We will compare the cell types present in the blood and the chemicals known to influence the human immune system before and after the drug is given, as well as measuring any changes in gene expression in white blood cells 4 and 24hrs after the drug is taken.

DETAILED DESCRIPTION:
Subjects will visit the University of Georgia (UGA) Clinical & Translation Research Unit (CTRU) twice on consecutive days and blood will be drawn from them. On the first occasion they will be weighed and will complete the consent process. They will have been randomly assigned to the test (Stromectol) or control (placebo) group, with 8 participants in the test group and 4 participants in the control group. Stromectol will be obtained from a medical supply distributor and a placebo will be obtained through the UGA School of Pharmacy. Drugs will be prescribed by Jonathan Murrow MD. They will be stored in their original packaging at room temperature in a drug locker in the lab at CTRU. Participants will be identified by number and allocated to groups using a block randomization protocol. Randomization and drug dispensation will be done by CTRU. Eighteen ml of blood will drawn in a fasting state and they will be administered 150 mcg/kg Stromectol or the equivalent number of placebo tablets immediately after blood is drawn. Participants will remain at CTRU for four hours after they take the drug, then another 15ml of blood will be drawn. On the second day they will attend CTRU at the same time and the third blood sample will be drawn 24 hrs after administration of the drug. On each occasion the drawn blood will be coded by CTRU staff prior to being collected by a member of the Department of Infectious Diseases and taken to the laboratory (Wildlife Health G0007) for the isolation of leukocyte populations (peripheral monocytes, lymphocytes and polymorphonuclear cells (PMNs)) and for the preparation of serum. Complete blood counts will also be carried out. Sera will be analyzed on the Luminex for cytokine/chemokine content. RNA will be isolated from the cell populations for RNASeq analysis.

ELIGIBILITY:
Inclusion Criteria:

* Weight over 110 pounds and under 185 pounds

Exclusion Criteria:

* Pregnancy or nursing mothers.
* Immunosuppressed individuals.
* Hypersensitivity to ivermectin, cellulose, starch, magnesium stearate, butylated hydroxyanisole, or citric acid powder (inert ingredients of Stromectol).
* Recent (last 3 years) travel to West or Central Africa, or any other country where onchocerciasis is present
* Hepatitis/HIV
* Currently taking warfarin
* Lactose intolerance (Lactose present in placebo)
* Currently taking Steroid medications (inhaled, oral or injection)
* Currently taking Barbiturates, Benzodiazepines such as Xanax or Klonopin, Valproic acid (Lithium), Calcium channel blockers, Statins (cholesterol medication)
* Liver or renal dysfunction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian J Wolstenholme, PhD, Principal Investigator — University of Georgia
Locations (1):
- University of Georgia, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wilson NE, Reaves BJ, Wolstenholme AJ. Lack of detectable short-term effects of a single dose of ivermectin on the human immune system. Parasit Vectors. 2021 Jun 5;14(1):304. doi: 10.1186/s13071-021-04810-6. PMID 34090504

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ivermectin | Control
Started | 8 | 4
Completed | 8 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ivermectin | Control | Total
Number analyzed (Participants) | 8 | 4 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 4 | 12
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 3 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 6 | 3 | 9
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 4 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: The Number of Cytokines Showing Statistically Significant Changes From Pre-treatment Levels Will be Recorded.
Description: Changes in serum levels of a panel of 41 cytokines will be compared to baseline levels using Luminex methods (HCYTOMAG-60K-PX41 kit from EMD Millipore). No pre-specified threshold was set for biological significance, and the number of cytokines showing a statistically significant (p=<0.05) change from time 0 for each group will be reported. The number of cytokines with significant changes is taken from a comparison of the mean levels in each of the groups, not at the level of individual participants.
Time Frame: Pre-treatment, 4 hours and 24 hours post-treatment
Population: Cytokines were measured in sera using the HCYTOMAG-60K-PX41 kit from EMD Millipore. The numbers reported are the number of cytokines with statistically significant changes ( p = <0.05) from pre-treatment levels.
Measure: Number; unit: Cytokines changed from t=0
Units Other Than Participants: Cytokines
Groups:
- Ivermectin 4hrs: Ivermectin will be administered once at 150mcg/kg, orally.
  Ivermectin: 150 mcg/kg ivermectin, by mouth. 4 hrs post-treatment
- Ivermectin 24 Hrs: Ivermectin will be administered once at 150mcg/kg, orally.
  Ivermectin: 150 mcg/kg ivermectin, by mouth.24 hrs post-treatment
- Control 4 Hrs: An oral placebo will be administered once
  Placebo: An oral placebo will be administered, once. Sera collected 4hrs post-treatment
- Control 24 Hrs: An oral placebo will be administered once
  Placebo: An oral placebo will be administered, once. Sera collected 24hrs post-treatment
Arm/Group | Ivermectin 4hrs | Ivermectin 24 Hrs | Control 4 Hrs | Control 24 Hrs
Number analyzed (Participants) | 8 | 8 | 4 | 4
Number analyzed (Cytokines) | 41 | 41 | 41 | 41
Cytokines changed from t=0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Ivermectin 4hrs vs Ivermectin 24 Hrs vs Control 4 Hrs vs Control 24 Hrs; All measurements were compared to the same group at t=0, that is before the drug or placebo was administered. We compared the expression levels for each transcript, using the mean levels in each group, not at the individual participant level; Test type: Other; We analyzed the changes is level for each cytokine between the groups. P value was adjusted for multiple comparisons and significance determined using the Holm-Sidak method. The threshold value for statistical significance for the mean value between groups was set at p =<0.05 for each cytokine measured. The number of cytokines that met this threshold is reported

2. Primary Outcome: Number of Transcripts in PBMC With Statistically Significant Changes From Pre-treatment Levels.
Description: Changes in expression levels of approximately 770 genes involved in innate immunity will be measured in peripheral blood mononuclear cells (PBMC) before and after treatment. The number of transcripts with significant changes is taken from a comparison of the mean levels in each of the groups, not at the individual participant level. No pre-determined threshold was set for the biological significance of these changes.
Time Frame: Pre-treatment, 4 hours and 24 hours post-treatment
Population: Levels of 770 messenger RNAs (mRNAs) were assayed in PBMC isolated from study participants using the Human Nanostring Myeloid cell panel.
Measure: Number; unit: Transcripts signicantly changed from t=0
Arm/Group | Ivermectin 4hrs | Ivermectin 24 Hrs | Control 4 Hrs | Control 24 Hrs
Number analyzed (Participants) | 8 | 8 | 4 | 4
Transcripts signicantly changed from t=0 | 0 | 0 | 10 | 0
Statistical Analysis 1: Comparison: Ivermectin 4hrs vs Ivermectin 24 Hrs vs Control 4 Hrs vs Control 24 Hrs; All measurements were compared to the same treated/control group at t=0, before the drug or placebo was administered. We compared the expression levels for each transcript, using the mean levels in each group, not at the individual participant level; Test type: Other; We compared the expression levels for each transcript, using the mean levels in each group, not at the individual participant level. The p-value for each transcript is adjusted for multiple comparisons across all 770 transcripts, using the Benjamini-Yekutieli method. The number reported is the number of transcripts where p=<0.05

3. Secondary Outcome: Complete Blood Counts (CBC)
Description: CBCs will be performed before treatment and 24 hrs later
Time Frame: Pre-treatment (0hrs), 24 hours
Measure: Mean (Standard Error); unit: Million cells/mL
Groups:
- Ivermectin 0 Hrs: Ivermectin will be administered once at 150mcg/kg, orally.
  Ivermectin: 150 mcg/kg ivermectin, by mouth. Blood collected at t=0
- Ivermectin 24 Hrs: Ivermectin will be administered once at 150mcg/kg, orally.
  Ivermectin: 150 mcg/kg ivermectin, by mouth.Blood collected 24 hrs post-treatment
- Control 0 Hrs: An oral placebo will be administered once
  Placebo: An oral placebo will be administered, once. Blood collected at t=0
- Control 24 Hrs: An oral placebo will be administered once
  Placebo: An oral placebo will be administered, once. Blood collected 24hrs post-treatment
Arm/Group | Ivermectin 0 Hrs | Ivermectin 24 Hrs | Control 0 Hrs | Control 24 Hrs
Number analyzed (Participants) | 8 | 8 | 4 | 4
Million cells/mL
  Neutrophils | 3.069 (0.353) | 3.341 (0.426) | 2.940 (0.18) | 3.358 (0.47)
  Lymphocytes | 1.753 (0.22) | 1.864 (0.151) | 1.833 (0.161) | 2.075 (0.175)
  Monocytes | 0.483 (0.045) | 0.403 (0.057) | 0.373 (0.04) | 0.375 (0.034)
  Eosinophils | 0.208 (0.055) | 0.205 (0.047) | 0.158 (0.015) | 0.170 (0.018)
  Basophils | 0.04 (0.008) | 0.046 (0.006) | 0.048 (0.008) | 0.048 (0.0005)
Statistical Analysis 1: Comparison: Ivermectin 0 Hrs vs Ivermectin 24 Hrs vs Control 0 Hrs vs Control 24 Hrs; Test type: Other; p < 0.05, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 1 day following administration of the drug/placebo
Arm/Group | Ivermectin | Control
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/4
Other Adverse Events (participants affected / at risk) | 1/8 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ivermectin (N=8) | Control (N=4)
Minor gastrointestinal upset (Gastrointestinal disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/94/NCT03459794/Prot_SAP_ICF_000.pdf